CLINICAL TRIAL: NCT04201444
Title: Usefulness of Hair Cortisol/Cortisone Concentrations for the Monitoring of Medical Treatment in Patients With Cushing's Disease
Brief Title: Hair Cortisol and Cushing's Disease
Acronym: HAIRCUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2018/60
Record Dates: First submitted 2019-09-04; First posted 2019-12-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Cushing Disease
Keywords: UFC; LNSC; Hair cortisol; medical treatment
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient group (Experimental)
  Interventions: Diagnostic Test: Patient group
- Remission control group (Active Comparator)
  Interventions: Diagnostic Test: Remission control group
- Bilateral surrenalectomy control group (Active Comparator)
  Interventions: Diagnostic Test: Bilateral surrenalectomy control group

INTERVENTIONS:
Diagnostic Test: Patient group — Patients with Cushing Disease (CD) receiving a medical treatment: n = 30 Plasmatic cortisol UFC Urine biocollection Salive biocollection
  Arms: Patient group
Diagnostic Test: Remission control group — Patients in remission of CD and having recovered a normal pituitary function for at least 12 months following pituitary surgery (normal UFC associated to: cortisol suppression following dexamethasone suppression test, or normal LNSC, or midnight serum cortisol < 200 nmol/L) n = 15 Plasmatic cortisol UFC Urine biocollection Salive biocollection Haircortisol
  Arms: Remission control group
Diagnostic Test: Bilateral surrenalectomy control group — Patients with previous CD, treated with bilateral adrenalectomy and receiving weight adjusted doses of hydrocortisone for at least 6 months. Last daily dose of Hydrocortisone should be administered no later than 5 pm. n = 15 Plasmatic cortisol UFC Urine biocollection Salive biocollection Haircortisol
  Arms: Bilateral surrenalectomy control group

SUMMARY:
The biochemical tools usable to assess the control of hypercortisolism in patients with Cushing's disease receiving medical treatments are debatable. The aim of the study is to compare the results of the measurement of cortisol and cortisone using high-performance liquid chromatography-tandem mass spectrometry (LC-MS/MS) in scalp hair (so called "Hair Cortisol") to that of 24h urinary free cortisol (UFC) and late night salivary cortisol (LNSC) for the monitoring of medical therapy in patients with Cushing's disease (CD).

DETAILED DESCRIPTION:
Selective surgical removal of the pituitary corticotroph adenoma is the ideal treatment of Cushing's disease. However, surgery may not be feasible or is unsuccessful in roughly 25% of patients. In addition, a recurrence of the disease is observed after a transient remission in 15 to 25% of patients. Several therapeutic alternatives are available, amongst which medical treatment is commonly used. Drugs that are available in France to control hypercortisolism target the pituitary adenoma secretion (pasireotide and cabergoline) or inhibit adrenal steroidogenesis (ketoconazole and metyrapone). Usual criteria to monitor the treatment and titrate the drug dosage include evaluation of relevant clinical endpoints and measurement of UFC. However, limitations of UFC for this purpose, include difficulties in obtaining a complete 24 urine collection and the fact that UFC assess only short-term cortisol in a disease characterized by high variability over time in the intensity of hypercortisolism. Elsewhere, a mild to moderate hypercortisolism may persist despite a normal UFC. Several groups, including ours, have shown that LNSC is useful tool to diagnose overt and mild hypercortisolism and may be more sensitive than UFC to diagnose mild hypercortisolism. Despite being more convenient to collect than 24h urine, LNSC also suffers from only measuring time-point cortisol. Rare studies have examined whether LNSC could be an adequate biomarker for monitoring response to medical therapy in patients with CD and its usefulness to monitor drug treatment in CD is yet unknown (one study comparing UFC to LNSC in CD patients treated with pasireotide-LAR has been presented but is not yet published). Accordingly, the 2015 guidelines of the endocrine society recommend future research to accurately monitor patients for their response to medical therapy to guide dose optimization. More recently, the measurement of salivary cortisone in 3 saliva samples (SCx3) drawn at approximately 8 hours intervals and starting at 7-8 am have been shown to be a reliable estimate of cortisol production over 24h in normal subjects. Whether this parameter could be used as a substitute of UFC in patients treated with anticortisolic drugs remains unstudied.

Hair cortisol concentration is a non-invasive way to measure cortisol exposure over much longer periods of time (weeks and months) than previously possible with samples of blood, saliva or urine. Several studies have shown that measurement of cortisol in a single scalp hair sample has a diagnostic accuracy for CS similar to currently used first-line tests and may also be used to identify overtreatment in patients receiving hydrocortisone replacement for adrenal insufficiency. To date, no data is available concerning hair Cortisol measurement in comparison with other usual biological tools in patients with CD receiving a medical treatment.

Since 2016, the departments of endocrine biology and clinical endocrinology of Bordeaux university hospital (CHU) have developed the measurement of cortisol and cortisone in scalp hair using LC-MS/MS and have established normative values using several cohorts of control patients.

The purpose of the study is to take advantage of the ability of hair cortisol to measure long-term cortisol exposure to assess the response to medical therapy in patients with CD. More specifically, the working hypothesis is that some patients with a normal UFC may still suffer from an occult mild hypercortisolism that will be identified only by hair cortisol. To study this hypothesis, the investigators will compare the results of hair cortisol to that multiple measurement of UFC, LNSC and SCx3 during a three-month period in patients with CD already treated with medical treatments and considered as "controlled" on the basis of previous UFC measurements.

ELIGIBILITY:
Inclusion Criteria:

In the three groups:

* Age > 18
* Cushing's disease medical history: histology confirming an ACTH staining adenoma, or ACTH-dependant Cushing syndrome with MRI confirmation of pituitary adenoma, or pituitary secretion of ACTH confirmed with petrosal sinus gradient
* Written informed consent
* Hair length ≥ 3 cm

In patient group:

* Persistent CD diagnosed on usual criteria in expert centers including overt hypercortisolism with at least 2 UFC > 1.5 N prior to the start of medical treatment
* Previous treatment with pasireotide, cabergoline, metyrapone, ketoconazole (alone or in association) AND hypercortisolism considered as controlled for at least 3 months based on 2 normal UFC.

In remission control group:

o Patients cured of CD and having recovered a normal pituitary function for at least 12 months following pituitary surgery (normal UFC associated to: cortisol suppression following dexamethasone suppression test, or normal LNSC, or midnight serum cortisol < 200 nmol/L)

In bilateral surrenalectomy control group:

o Patients with previous CD, treated with bilateral adrenalectomy and receiving weight adjusted doses of hydrocortisone for at least 6 months. Last daily dose of Hydrocortisone should be administered no later than 5 pm.

Exclusion Criteria:

In the three groups:

* Renal Failure (Cl < 30 mL/min)
* Non-compliant patients
* Hair length < 3 cm
* Severe depression and psychosis
* Drug addiction and active alcoholism
* Myocardial infarction or cerebrovascular accident < 3 months
* Intense physical activity (marathon runner)
* Night-shifters
* Obesity with BMI > 35 kg/m2
* Type 1 diabetes
* Type 2 diabetes with HbA1C > 9 %

In patient group:

* Patients receiving mifepristone and/or mitotane
* Patients treated with anticortisolic agents during the titration process
* Patients requiring additional hydrocortisone supplementation or exogenous corticosteroids
* Pituitary radiotherapy < 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Evaluate cortisol chronic tissue impregnation | 3 months after inclusion day
  Hypercortisolism will be controlled using 3 cm scalp hair sample in which Hair Cortisol will be measured in patients with Cushing Disease (CD) receiving a medical treatment.

SECONDARY OUTCOMES:
Evaluate Hair Cortisol (Hcort) measure for Cushing Disease control | 3 months after inclusion day
  Compare Hair Cortisol to UFC (Urinary Free Cortisol), LNSC (late night salivary cortisol) and SC (salivary cortisone) in patients with CD receiving a medical treatment.
Compare cortisol tissue impregnation thanks to Hair Cortisol measurements in patients with CD receiving a medical treatment and patients control | 3 months after inclusion day
  Compare the results of Hair Cortisol measurements in patients with CD receiving a medical treatment and patients treated with weight-adjusted hydrocortisone replacement doses after bilateral adrenalectomy
Compare cortisol tissue impregnation thanks to Hair Cortisol measurements in patients cured from CD and patient with bilateral adrenalectomy | 3 months after inclusion day
  Compare the results of Hair Cortisol measurements in patients cured from CD and patients with bilateral adrenalectomy
Evaluate Hair Cortisol intra-individual variability | At day 0 and day 90
  Evaluate the dosage of within-patient variability of Hair Cortisol for patients with CD receiving a medical treatment and control groups : patients cured from CD and patients with bilateral adrenalectomy
Evaluate UFC intra-individual variability | 3 months after inclusion day
  Assess the within-patient variability of UFC in patients with CD receiving a medical treatment
Satisfaction assessed by Cushing's QOL | 3 months after inclusion day
  Correlate a quality of life assessment with the results of Hair Cortisol, UFC and LNSC thanks to QOL questionnaire : cushing's QOL.
Evaluate LNSC intra-individual variability | 3 months after inclusion day
  Evaluate the dosage of within-patient variability of LNSC in patients with CD receiving a medical treatment
Evaluate SC intra-individual variability | 3 months after inclusion day
  Evaluate the dosage of within-patient variability of SC in patients with CD receiving a medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Antoine TABARIN, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - Service d'Endocrinologie - CHU Caen, Caen
  - Service d'endocrinologie - HCL, Lyon
  - Service d'Endocrinologie, Diabète et Maladies Métaboliques - APHM, Marseille
  - CIC d'Endocrinologie, Maladies Métaboliques et Nutrition - CHU de Nantes, Nantes
  - Service d'Endocrinologie - APHP Cochin, Paris
  - Service d'Endocrinologie et des Maladies de la Reproduction - APHP Bicêtre, Paris
  - Service d'endocirnologie, diabète, nutrition, Hôpital Haut Lévêque - CHU de Bordeaux, Pessac

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohammedi K, Bertherat J, Raverot G, Drui D, Reznik Y, Castinetti F, Chanson P, Fafin M, Brossaud J, Tabarin A. Evidence of Persistent Mild Hypercortisolism in Patients Medically Treated for Cushing Disease: the Haircush Study. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e963-e970. doi: 10.1210/clinem/dgad251. PMID 37144820